CLINICAL TRIAL: NCT04381520
Title: Heat-sensitive Moxibustion Self-administration in Patients in the Community With Primary Hypertension: Protocol for a Multi-center, Pragmatic, Non-randomized Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangxi University of Traditional Chinese Medicine (Other)
Collaborators: Nangang community healthcare center (Nanchang city, Jiangxi province, China) (Unknown); Honggutan community healthcare center (Nanchang city, Jiangxi province, China) (Unknown); Shengmi community healthcare center (Nanchang city, Jiangxi province, China) (Unknown); Gaofu town community healthcare center (Fu Zhou city, Jiangxi province, China) (Unknown)
Responsible Party: Principal Investigator, Xu Zhou, Associate professor, Jiangxi University of Traditional Chinese Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JXUTCM-Mox-01
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Primary Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Antihypertensive Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heat-sensitive moxibustion plus antihypertensive drugs (Experimental)
  Interventions: Other: Heat-sensitive moxibustion plus antihypertensive drugs
- Antihypertensive drugs (Active Comparator)
  Interventions: Drug: Antihypertensive drugs

INTERVENTIONS:
Other: Heat-sensitive moxibustion plus antihypertensive drugs — In this arm, patients will administer heat-sensitive moxibustion by themselves or by the help of their family after professional training. Patients will maintain their original antihypertensive drugs. The periods of treatment and follow-up will be one year.
  Arms: Heat-sensitive moxibustion plus antihypertensive drugs
Drug: Antihypertensive drugs — In this arm, patients will maintain their original antihypertensive drugs. The periods of treatment and follow-up will be one year.
  Arms: Antihypertensive drugs

SUMMARY:
Heat-sensitive moxibustion is considered to be effective for primary hypertension in hospital setting. This study aims to investigate whether heat-sensitive moxibustion self-administration is effective for lowering blood pressure and improving quality of life for patients with primary hypertension in community setting using a multicenter, prospective, non-randomized study design

DETAILED DESCRIPTION:
Primary hypertension is a global health issue with high incidence; it affected approximately 1.13 billion people worldwide and directly or indirectly causing an 10.4 million of death yearly. The routine drugs for primary hypertension are limited by adverse effects and expensive costs. Therefore, complementary and alternative medicine with good efficacy and safety and low expenditure is still needed for primary hypertension, especially in poverty-stricken areas.

Heat-sensitive moxibustion is an innovative therapy developed on the basis of traditional moxibustion. Compared with traditional moxibustion, heat-sensitive moxibustion advocates finding heat-sensitive acupoints where patients have special reactions to moxibustion heat, including diathermy, heat transfer, soreness, etc. The application of moxibustion on heat-sensitive acupoints (i.e., heat-sensitive moxibustion) has been shown to be more effective to traditional moxibustion for many diseases, including primary hypertension. Moreover, compared with acupuncture, heat-sensitive moxibustion has a main advantage that moxibustion does not require professional qualifications and patients can self-administer moxibustion after professional training. However, the current evidence is generated only from hospital settings. Therefore, this study is specifically designed to investigate whether heat-sensitive moxibustion self-administration is an effective intervention for lowering blood pressure and improving quality of life for patients with primary hypertension in community setting.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria of primary hypertension
2. 18 to 70 years old
3. Sign the informed consent

Exclusion Criteria:

1. Secondary hypertension caused by kidney disease, macrovascular disease, pregnancy, endocrine disease, brain disease, drug-induced factors, etc.
2. Allergic to moxibustion equipment, moxa smoke or moxa
3. Pregnancy or lactation
4. A history of serious cardiovascular and cerebrovascular events such as cerebrovascular accidents and myocardial infarction
5. Complicated by liver and kidney dysfunction indicated by total bilirubin, alanine aminotransferase, aspartate aminotransferase, or blood creatinine are more than 2 times upper limit of normal value
6. Complicated by malignant tumors
7. Complicated by major mental disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 767 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in systolic blood pressure (mmHg) | Baseline, 6 months, and 12 months
Changes in diastolic blood pressure (mmHg) | Baseline, 6 months, and 12 months
Changes in dose of antihypertensive drugs | Baseline, 6 months, and 12 months
  Measured by percentage changes

SECONDARY OUTCOMES:
Total score of quality of life assessed by a validated patient-reported outcome scale | Baseline, 6 months, and 12 months
  Including 27 items and assessing impacts of hypertension on on the three dimensions, physical (18 items), psychological (4 items) and family-social (5 items). Each item is classified as five grades (0-4 points). The total score ranges from 0 to 108 points. A higher score indicates a worse quality of life.
Physical score of quality of life assessed by a validated patient-reported outcome scale | Baseline, 6 months, and 12 months
  Including 18 items. Each item is classified as five grades (0-4 points). The total score ranges from 0 to 72 points. A higher score indicates a worse quality of life.
Psychological score of quality of life assessed by a validated patient-reported outcome scale | Baseline, 6 months, and 12 months
  Including 4 items. Each item is classified as five grades (0-4 points). The total score ranges from 0 to 16 points. A higher score indicates a worse quality of life.
Family-social score of quality of life assessed by a validated patient-reported outcome scale | Baseline, 6 months, and 12 months
  Including 5 items. Each item is classified as five grades (0-4 points). The total score ranges from 0 to 20 points. A higher score indicates a worse quality of life.
Changes in fasting blood glucose (mg/dl) | Baseline, 6 months, and 12 months
Changes in glycated hemoglobin (%) | Baseline, 6 months, and 12 months
Changes in total cholesterol (mg/dl) | Baseline, 6 months, and 12 months
Changes in triglycerides (mg/dl) | Baseline, 6 months, and 12 months
Changes in low density lipoprotein cholesterol (mg/dl) | Baseline, 6 months, and 12 months
Changes in high density lipoprotein cholesterol (mg/dl) | Baseline, 6 months, and 12 months
Changes in urinary albumin (g/l) | Baseline, 6 months, and 12 months
Changes in serum creatinine (μmol/l) | Baseline, 6 months, and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangxi University of Traditional Chinese Medicine, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) of this study will be available from the principal investigator on reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After all results are published.

REFERENCES:
- [Derived] Zhou X, Wu Q, Zhang G, Wang Y, Li S, Wang B, Chen Z, Zhu W, Wang F, Gan C. Heat-sensitive moxibustion self-administration in patients in the community with primary hypertension: A protocol for a multi-center, pragmatic, non-randomized trial. Medicine (Baltimore). 2020 Sep 18;99(38):e22230. doi: 10.1097/MD.0000000000022230. PMID 32957364